CLINICAL TRIAL: NCT01304511
Title: Post-Marketing Surveillance Orgalutran (Ganirelix)®
Brief Title: Post-Marketing Surveillance of the Safety and Efficacy of Orgalutran (Ganirelix)®
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P08198
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Fertilization in Vitro
MeSH Terms: interventions — ganirelix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Treated: Women undergoing controlled ovarian COH for ART
  Interventions: Drug: Orgalutran

INTERVENTIONS:
Drug: Orgalutran
  Other Names: Ganirelix®

SUMMARY:
The purpose of this post-marketing surveillance is to identify problems and questions regarding the safety and efficacy of Orgalutran (Ganirelix)® when used for the prevention of premature luteinizing hormone (LH) surges in women undergoing controlled ovarian hyperstimulation (COH) for assisted reproduction techniques (ART).

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing COH for ART

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Hypersensitivity to gonadotropin-releasing hormone (GnRH) or any other GnRH analogue
* Moderate or severe impairment of renal or hepatic function
* Pregnancy or lactation

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing COH for ART
Sampling Method: Non-Probability Sample
Enrollment: 711 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes by COH based on Per stage approach | Baseline to End of Study
Number of Serious Adverse Events | Baseline to End of Study
Number of Unlabeled (Unexpected) Adverse Drug Reactions | Baseline to End of Study
Number of Labeled Adverse Drug Reactions | Baseline to End of Study
Number of Non-serious Adverse Events | Baseline to End of Study
Number of Adverse events by drug misuse/abuse or drug-drug interaction | Baseline to End of Study